CLINICAL TRIAL: NCT00345800
Title: Single Center, Therapeutic Exploratory Clinical Trial to Evaluate the Safety of Sodium Oxybate (Xyrem) 500 mg/mL Oral Solution on Potential Endocrine Changes at Currently Labeled Therapeutic Dose Regimens (4.5 - 9 g/Day Divided Into Two Equal Doses) During 12 Weeks of Treatment of Cataplexy in Adult Patients With Narcolepsy.
Brief Title: Exploratory Clinical Study to Evaluate Sodium Oxybate (Xyrem) on Potential Endocrine Changes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C00301; 2005-004417-15 (EudraCT Number)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-02

CONDITIONS: Narcolepsy With Cataplexy
Keywords: Endocrine Evaluation cataplexy; sodium oxybate (xyrem)
MeSH Terms: conditions — Narcolepsy | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Oxybate (Experimental): * Active Substance: Sodium Oxybate
  * Pharmaceutical form: Oral Solution
  * Concentration: 500 mg/mL oral solution from 4.5 to 9 g/day divided into two equal doses during 12 weeks
  * Route of administration: Oral
  Interventions: Drug: Sodium Oxybate (Xyrem)

INTERVENTIONS:
Drug: Sodium Oxybate (Xyrem) — * Active Substance: Sodium Oxybate
  * Pharmaceutical form: Oral Solution
  * Concentration: 500 mg/mL oral solution from 4.5 to 9 g/day divided into two equal doses during 12 weeks
  * Route of administration: Oral
  Other Names: Xyrem

SUMMARY:
To monitor for endocrine changes in response to treatment of cataplexy with Xyrem, to focus on the hypothalamic pituitary axis and to confirm the safety of Xyrem on potential endocrine changes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Narcoleptic patients with cataplexy

Exclusion Criteria:

* Subjects not diagnosed with narcolepsy with cataplexy

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-04-10 (Actual); Primary Completion 2008-01-22 (Actual); Study Completion 2008-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (1):
- Liège, Belgium

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center, therapeutic, exploratory study started to enroll subjects in April 2006.
Pre-assignment Details: Participant Flow refers to the Intention-to-Treat (ITT) population consisting of the 25 subjects enrolled in the study who took at least 1 dose of study medication.
Groups:
- Sodium Oxybate: Active Substance: Sodium Oxybate Pharmaceutical form: Oral Solution Concentration: 500 mg/mL oral solution from 4.5 to 9 g/day divided into two equal doses during 12 weeks Route of administration: Oral
Period: Overall Study
Arm/Group | Sodium Oxybate
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-to-Treat (ITT) population consisting of the 25 subjects enrolled in the study who took at least 1 dose of study medication.
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 23
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.99 (13.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: The Insulin-like Growth Factor 1 (IGF-1) Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of IGF-1 was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: Intention-to-Treat (ITT) population consisting of the 25 subjects enrolled in the study who took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ng/mL | 207.4 (86.5)

2. Primary Outcome: The Insulin-like Growth Factor 1 (IGF-1) Measured in Fasting Conditions After 1 Month of Treatment (Visit 3)
Description: An assay of IGF-1 was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: After 1 month of treatment (Visit 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ng/mL | 200.4 (77.7)

3. Primary Outcome: The Insulin-like Growth Factor 1 (IGF-1) Measured in Fasting Conditions After 3 Months of Treatment (Visit 4)
Description: An assay of IGF-1 was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: After 3 months of treatment (Visit 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ng/mL | 210.2 (90.3)

4. Secondary Outcome: The Circadian Rhythm of the Growth Hormone (GH) Measured at Baseline (Visit 2)
Description: Blood was sampled at Baseline (Visit 2) at bedtime 10:00 pm and 1, 2, 4, 8, 12, 16, and 20 hours after bedtime for assaying GH.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ng/mL
  Bed time | 1.821 (4.844)
  1h | 1.225 (2.895)
  2h | 1.408 (1.656)
  4h | 1.236 (1.904)
  8h | 0.576 (0.632)
  12h | 0.293 (0.310)
  16h | 0.309 (0.282)
  20h | 0.313 (0.362)

5. Secondary Outcome: The Circadian Rhythm of the Growth Hormone (GH) Measured at Visit 3
Description: Blood was sampled predose and 1, 2, 4, 8, 12, 16, and 20 hours postdose at Visit 3 for assaying GH.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ng/mL
  Pre-dose | 2.432 (7.118)
  1h | 5.914 (9.743)
  2h | 5.238 (8.557)
  4h | 3.018 (4.332)
  8h | 0.256 (0.326)
  12h | 0.308 (0.664)
  16h | 0.460 (0.767)
  20h | 0.306 (0.342)

6. Secondary Outcome: The Circadian Rhythm of the Growth Hormone (GH) Measured at Visit 4
Description: Blood was sampled predose and 1, 2, 4, 8, 12, 16, and 20 hours postdose at Visit 4 for assaying GH.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ng/mL
  Pre-dose | 0.816 (1.372)
  1h | 3.804 (3.173)
  2h | 3.864 (5.731)
  4h | 2.712 (3.178)
  8h | 0.224 (0.292)
  12h | 0.420 (1.355)
  16h | 0.296 (0.491)
  20h | 0.244 (0.390)

7. Secondary Outcome: Cortisol Measured at Baseline (Visit 2)
Description: Blood was sampled at Baseline (Visit 2) at bedtime 10:00 pm and 1, 2, 4, 8, 12, 16, and 20 hours after bedtime for assaying cortisol.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ug/L
  Bed time | 42.21 (28.53)
  1h | 27.91 (17.09)
  2h | 22.80 (14.54)
  4h | 36.06 (28.46)
  8h | 115.79 (52.33)
  12h | 143.39 (70.67)
  16h | 90.84 (34.83)
  20h | 68.48 (40.77)

8. Secondary Outcome: Cortisol Measured at Visit 3
Description: Blood was sampled predose and and 1, 2, 4, 8, 12, 16, and 20 hours postdose at Visit 3 for assaying cortisol.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ug/L
  Pre-dose | 35.84 (27.83)
  1h | 24.75 (18.20)
  2h | 34.62 (31.93)
  4h | 44.28 (36.64)
  8h | 95.61 (57.14)
  12h | 130.21 (61.28)
  16h | 77.33 (32.93)
  20h | 70.49 (33.71)

9. Secondary Outcome: Cortisol Measured at Visit 4
Description: Blood was sampled predose and 1, 2, 4, 8, 12, 16, and 20 hours postdose at Visit 4 for assaying cortisol.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ug/L
  Pre-dose | 34.46 (24.85)
  1h | 25.61 (19.06)
  2h | 30.06 (24.40)
  4h | 45.27 (35.65)
  8h | 113.84 (71.18)
  12h | 146.33 (64.42)
  16h | 92.48 (30.94)
  20h | 75.55 (38.01)

10. Secondary Outcome: The Adrenocorticotropic Hormone (ACTH) Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of ACTH was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
pg/mL | 65.6 (46.7)

11. Secondary Outcome: The Adrenocorticotropic Hormone (ACTH) Measured in Fasting Conditions at Visit 3
Description: An assay of ACTH was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
pg/mL | 62.8 (37.9)

12. Secondary Outcome: The Adrenocorticotropic Hormone (ACTH) Measured in Fasting Conditions at Visit 4
Description: An assay of ACTH was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
pg/mL | 54.8 (27.3)

13. Secondary Outcome: The Dehydroepiandrosterone Sulfate (DHEA-S) Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of DHEA-S was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ug/L | 1988.2 (1283.3)

14. Secondary Outcome: The Dehydroepiandrosterone Sulfate (DHEA-S) Measured in Fasting Conditions at Visit 3
Description: An assay of DHEA-S was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ug/L | 2200.9 (1517.5)

15. Secondary Outcome: The Dehydroepiandrosterone Sulfate (DHEA-S) Measured in Fasting Conditions at Visit 4
Description: An assay of DHEA-S was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
ug/L | 2130.7 (1450.4)

16. Secondary Outcome: The Prolactin Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of prolactin was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mUI/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mUI/L | 356.8 (185.9)

17. Secondary Outcome: The Prolactin Measured in Fasting Conditions at Visit 3
Description: An assay of prolactin was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mUI/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mUI/L | 280.0 (162.8)

18. Secondary Outcome: The Prolactin Measured in Fasting Conditions at Visit 4
Description: An assay of prolactin was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mUI/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mUI/L | 258.4 (113.6)

19. Secondary Outcome: The Thyroid Stimulating Hormone (TSH) Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of TSH was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
uU/mL | 1.366 (0.622)

20. Secondary Outcome: The Thyroid Stimulating Hormone (TSH) Measured in Fasting Conditions at Visit 3
Description: An assay of TSH was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
uU/mL | 1.292 (0.599)

21. Secondary Outcome: The Thyroid Stimulating Hormone (TSH) Measured in Fasting Conditions at Visit 4
Description: An assay of TSH was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
uU/mL | 1.425 (0.818)

22. Secondary Outcome: The Total Thyroxin (T4) Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of T4 was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
pg/mL | 11.34 (1.68)

23. Secondary Outcome: The Total Thyroxin (T4) Measured in Fasting Conditions at Visit 3
Description: An assay of T4 was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
pg/mL | 11.47 (2.10)

24. Secondary Outcome: The Total Thyroxin (T4) Measured in Fasting Conditions at Visit 4
Description: An assay of T4 was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
pg/mL | 11.65 (1.78)

25. Secondary Outcome: The Osmolality Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of osmolality was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mosm/kg
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mosm/kg | 291.6 (4.5)

26. Secondary Outcome: The Osmolality Measured in Fasting Conditions at Visit 3
Description: An assay of osmolality was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mosm/kg
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mosm/kg | 292.2 (4.9)

27. Secondary Outcome: The Osmolality Measured in Fasting Conditions at Visit 4
Description: An assay of osmolality was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mosm/kg
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mosm/kg | 292.1 (5.5)

28. Secondary Outcome: Electrolytes (Na, K, Ca) Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of electrolytes was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mmol/L
  Na (Sodium in mmol/L) | 141.4 (1.9)
  K (Potassium in mmol/L) | 3.88 (0.21)
  Ca (Calcium in mmol/L) | 2.257 (0.084)

29. Secondary Outcome: The Electrolyte Phosphate (P) Measured in Fasting Conditions at Baseline (Visit 2)
Description: An assay of electrolytes was done from blood sampled about 10 hours after bedtime on Visit 2.
Time Frame: Baseline (Visit 2) - approximately 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mg/L | 34.4 (6.0)

30. Secondary Outcome: Electrolytes (Na, K, Ca) Measured in Fasting Conditions at Visit 3
Description: An assay of electrolytes was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mmol/L
  Na (Sodium in mmol/L) | 141.9 (2.1)
  K (Potassium in mmol/L) | 3.90 (0.25)
  Ca (Calcium in mmol/L) | 2.334 (0.071)

31. Secondary Outcome: The Electrolyte Phosphate (P) Measured in Fasting Conditions at Visit 3
Description: An assay of electrolytes was done from blood sampled about 10 hours postdose on Visit 3.
Time Frame: Visit 3 (approximately 1 month)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mg/L | 34.2 (4.5)

32. Secondary Outcome: Electrolytes (Na, K, Ca) Measured in Fasting Conditions at Visit 4
Description: An assay of electrolytes was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mmol/L
  Na (Sodium in mmol/L) | 141.2 (1.9)
  K (Potassium in mmol/L) | 3.80 (0.27)
  Ca (Calcium in mmol/L) | 2.290 (0.063)

33. Secondary Outcome: The Electrolyte Phosphate (P) Measured in Fasting Conditions at Visit 4
Description: An assay of electrolytes was done from blood sampled about 10 hours postdose on Visit 4.
Time Frame: Visit 4 (approximately 3 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
mg/L | 35.0 (3.5)

34. Secondary Outcome: The Number of Patients Reporting at Least One Adverse Event (AE) During the Course of the Study
Description: An AE was classified as a treatment-emergent AE (TEAE) if its onset date and time was on or after the first study drug administration. Number of subjects with at least one TEAE is reported below.
Time Frame: Visit 1 through the end of the study (approximately 4 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
Participants | 20

35. Secondary Outcome: The Number of Patient Withdrawal Due to Adverse Events (AEs) During the Course of the Study
Description: An AE was classified as a treatment-emergent AE (TEAE) if its onset date and time was on or after the first study drug administration. Number of subjects with TEAE that led to temporarily discontinuation of study drug is reported below.
Time Frame: Visit 1 through the end of the study (approximately 4 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
Participants | 1

36. Secondary Outcome: The Number of Patients Reporting at Least One Serious Adverse Event (SAE) During the Course of the Study
Description: A Serious Adverse Event is any untoward medical occurrence that at any dose • results in death, • is life threatening, • requires in-patient hospitalization or prolongation of existing hospitalization, • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect
Time Frame: Visit 1 through the end of the study (approximately 4 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 25
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Visit 1 through the end of the study (approximately 4 months).
Description: Adverse Events refer to the Safety Population which is identical to the Intention-to-Treat (ITT) population consisting of the 25 subjects enrolled in the study who took at least 1 dose of study medication.
Arm/Group | Sodium Oxybate
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oxybate (N=25)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oxybate (N=25)
Nausea (Gastrointestinal disorders) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (4)
Headache (Nervous system disorders) | 6 (8)
Dizziness (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days